CLINICAL TRIAL: NCT06139003
Title: Evaluation of Digital Versus Conventional Techniques for Construction of Mandibular Implant Retained Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A02060922
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Occlusal Wear of Teeth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3d Printed implant overdenture (Experimental): patients will receive maxillary CD and mandibular 2-implant retained overdenture over locator attachment constructed by digital technique.
  Interventions: Device: 3d Printed implant
- Conventionally constructed implant overdenture (Experimental): patients will receive maxillary CD and mandibular 2-implant retained overdenture over locator attachment constructed by conventional technique.
  Interventions: Device: Conventionally constructed implant

INTERVENTIONS:
Device: 3d Printed implant — Occlusal stability was evaluated using occlusense device by charting amount and distribution of force over dental arch in percentage
  Arms: 3d Printed implant overdenture
Device: Conventionally constructed implant — Occlusal stability was evaluated using occlusense device by charting amount and distribution of force over dental arch in percentage
  Arms: Conventionally constructed implant overdenture

SUMMARY:
The aim of this study is to evaluate of two different construction techniques (digital and conventional techniques) for two implant retained complete mandibular overdenture regarding:

1. Digital occlusion stability detection: evaluated by using OccluSense.

Evaluation was done in the following evaluation period:

T0: Immediately after over denture insertion. T6: 6 months after over denture insertion. T12: 12 months after over denture insertion.

DETAILED DESCRIPTION:
Patient selection and study design:

Six patients who required complete denture were selected from the diagnostic clinic of Prosthodontic Department, Faculty of Dentistry, Mansoura University. All patients were informed about the procedures that was done and a written consent form of ethical committee. All patients had the right to withdraw from the study at any time.

Patients Grouping:

Patients were divided in to 2 equal groups:

Group (I): 3 patients received maxillary CD and mandibular 2-implant retained overdenture constructed by digital technique.

Group (II): 3 patients received maxillary CD and mandibular 2-implant retained overdenture constructed by conventional technique.

Surgical phase procedures:

1. Preoperative investigations of the patient were done that included the blood profile (hemoglobin, complete blood (cell) count, bleeding time, clotting time, random blood sugar).
2. Preoperative assessment of mandibular bone was done radiographically by cone beam computerized tomography (CBCT).
3. Each patient received two dental implants in the canine area bilaterally.
4. All implants were placed according to the flapless protocol.
5. A customized surgical stent fabricated according to the preoperative computer based 3D plan and used during the surgical procedure to ensure accurate implant position and angulation.
6. A small round bur (or Guide drill) the first drill used to make a hole of 1-2 mm deep to create a start point for the pilot drill.
7. The pilot drill is the first twist drill used to create the osteotomy up to the desired length.
8. The drills should be repeatedly pumped in and out of the osteotomy to expose the bone debris to the water coolants for clearing.
9. A guide pin should be placed in the prepared site to check alignment and parallelism.
10. Subsequent drills were used in the same way as the pilot drill to enlarge the osteotomy to the desired depth.
11. Profile drills or countersink drills were used to widen the crestal part of the osteotomy to allow the next drill into the osteotomy and to allow the placement of the cover screw without any bony interference.
12. Osteotomy was performed through the sleeves of the surgical stent and the implants were placed by hand using a torque wrench (35-45 Ncm) through the sleeves. the implant placed 0.5 mm slightly subcrestal, and cover screws were secured using Hex driver.
13. The dentures were molded to not interfere with the peri-implant tissues and reduce occlusal forces on the implant.

After 3 months of osteointegration period, the implants were exposed, the cover screw was removed and the two healing abutments were screwed into the fixture using their driver for 7 to 10 days.

Each patient received maxillary complete denture against mandibular 2- implant retained complete overdenture with two different construction techniques.

The clinical procedures in the respective visits are described below:

Steps of conventional complete overdenture construction:

1. For each patient in group two, preliminary maxillary and mandibular impressions were made using irreversible hydrocolloid impression material and stock impression trays.
2. on custom trays border molding performed by using a thermoplastic compound green sticks.
3. The maxillary definitive impressions were made by using a zinc oxide impression material.

6. The mandibular definitive impressions were made by direct impression technique with the aid of impression post and laboratory analogue.

7. Models were poured with implant analogues; the definitive locator attachment was screwed.

8. Fabrication of maxillary and mandibular record blocks were done and the labial fullness was established, occlusal plane, and occlusal vertical dimension was recorded and the reference lines (midline and canine line) was marked on the wax rims.

9. Centric jaw relation was registered. Using face bow, upper cast mounted and then centric relation recorded.

10. Selection of teeth was done by using the readymade artificial acrylic teeth with lingualized occlusal scheme. And setting of teeth was done with bilateral balanced occlusion.

11. Try-in, processing, finish and polish of the dentures were done.

Digital complete overdenture construction:

1. For each patient in group one, preliminary maxillary and mandibular impressions and poured with dental stone in casts and custom trays were fabricated.
2. Border molding performed. The maxillary and mandibular definitive impressions were made.
3. Models were poured with implant analogues; the definitive locator attachment was screwed.
4. Scanning for the model was done to achieve 3D virtual image to the models.
5. Fabrication of maxillary and mandibular record blocks were done and the labial fullness was established, occlusal plane, and occlusal vertical dimension was recorded and the reference lines (midline and canine line) marked on the wax rims and the resultant data was scanned.
6. The file of this master scan in STL format transmitted to the CADCAM complete denture provider using a purpose-built software program.
7. The anatomic landmarks identified, and the peripheral limits marked on a virtual model in the design software, which then was served to design the definitive denture base.
8. A virtual tooth arrangement was generated for a digital preview.
9. The digital preview was evaluated and modified if necessary.
10. Transfer data to a CAM software program, the prostheses printed, finished and polished.

Insertion the prosthesis into the patient's mouth and have them bit down until the resin has cured. Remove the prostheses and trim the excess resin. The prosthesis delivered and patient instructed about the aftercare and recall schedule steps.

Evaluation

Digital occlusal stability detection:

Group I and group II subjected to test by utilization of the Digital Occlusal Analyzer System (OccluSense). The occlusal forces distribution, extent and time sequence can then have recorded: Immediately, 6 and 12 months after denture use.

ELIGIBILITY:
Inclusion Criteria:

* healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis.
* Completely edentulous jaws for at least 1 year.
* The angle's class I maxillomandibular relationship and have upper and lower completely edentulous arches.
* Residual alveolar ridges covered with healthy firm mucosa.
* All included patients' sufficient available length and width of mandibular bone to accommodate conventional implant. (At least 5 mm buccolingual width and 12 mm vertical height of bone).

Exclusion Criteria:

* Patients with systemic diseases that contraindicate implant placement such as hematologic diseases
* metabolic diseases related to bone resorption such as uncontrolled diabetics or osteoporosis will be also excluded
* History of para-functional habits (Bruxism, clenching), smoking and alcoholism.
* History of radiation therapy in the head and neck region.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
occlusal stability | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Using occlusense device to determine distribution of occlusal forces over anterior and posterior areas, right and left side through chart representing areas of occlusal contact
Occlusal analysis | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Group I and group II will be subjected to test by utilization of the Digital Occlusal Analyzer System (OccluSense) then amount of occlusal force over each unit presented in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady, MD, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali AEA, Habib A, Shady M. Digital versus conventional techniques for construction of mandibular implant retained overdenture. BMC Oral Health. 2025 May 5;25(1):686. doi: 10.1186/s12903-025-05918-2. PMID 40325470